CLINICAL TRIAL: NCT06972329
Title: Cerebral Near Infrared Spectroscopy in Out-of-Hospital Cardiac Arrest and Neurological Prognosis
Acronym: NISOHCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, JAEGER Deborah, Coordinating Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022PI126; 2025-A00903-46 (Other: ANSM)
Record Dates: First submitted 2025-04-17; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: Out-of-hospital cardiac arrest; Cerebral Near infrared spectroscopy (NIRSc)
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Out-of-hospital cardiac arrest (OHCA) study cohort with Cerebral Near infrared spectroscopy (NIRSc).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cerebral Near infrared spectroscopy (NIRSc) group (Experimental): The use of cerebral Near infrared spectroscopy to predict the neurological prognosis of patients treated for out-of-hospital cardiac arrest.
  Interventions: Other: Cerebral Near infrared spectroscopy (NIRSc).

INTERVENTIONS:
Other: Cerebral Near infrared spectroscopy (NIRSc). — Continuous cerebral near-infrared spectroscopy (NIRSc) during resuscitation in a patient treated for out-of-hospital cardiac arrest (OHCA).

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) prognosis remains poor : 7% of patients surviving without neurological impairment.

65% of patients dying after hospital admission were neurologically impaired. When treating a patient with CA, neurological outcome remains extremely difficult to predict, especially in the pre-hospital setting. Practitioners have very little objective information to help them with neuropronostication.

Although an EtCO2 level of < 10 mmHg is associated with a poor neurological prognosis, European recommendations point out that this data alone is not currently sufficient to predict a patient's prognosis or to make a decision to stop resuscitation. Current recommendations do not suggest any other objective parameter during resuscitation for neuropronostication of patients with out-of-hospital cardiac arrest.

Cerebral tissue oxygen saturation (rSO2) is measured using the near infrared spectrometry (NIRS) technique. Cerebral NIRS (cNIRS) enables non-invasive measurement of changes in cerebral oximetry during the management of a cardiac arrest (CA).

Various clinical studies conducted over the last ten years have demonstrated that there is a probable link between cNIRS levels during resuscitation and return of spontaneous circulation (ROSC), but a clear threshold value has not been defined.

The aim of the NISOHCA study is to confirm that a 40% threshold of cNIRS in the pre-hospital setting for OHCA can specifically predict survival with good neurological outcome at D90 .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Non-traumatic out-of-hospital cardiac arrest witnessed and managed by the mobile emergency unit (SMUR).

Exclusion Criteria:

* Scalp/cranial or facial injury preventing the placement of electrodes for NIRS measurement.
* Spontaneous cardiac activity upon the arrival of the SMUR.
* Decision by the SMUR physician not to initiate specialized resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Cerebral Performance Category (CPC) | Day 90
  Specificity of predicting a 90-D survival with a good neurological outcome with a mean c-NIRS > 40% during Cardiopulmonary Resuscitation (CPR). Cerebral Performance Category (CPC) of 1 to 5. CPC 1: Complete recovery without neurological impairment or conscious with minor impairment. CPC 5: Deceased or brain dead.

SECONDARY OUTCOMES:
Cerebral Performance Category (CPC) | Day 90
  Determine the probability of observing a poor neurological prognosis at 90 days if the average cerebral NIRS (NIRSc) is below 40% during resuscitation.
  Determine the probability of observing a good neurological prognosis at 90 days if the average cerebral NIRS (NIRSc) is greater than or equal to 40% during resuscitation.
  Identify the most appropriate NIRSc threshold to predict a good neurological prognosis at 90 days.
  Build a multi-marker model for neurological prognosis including NIRSc.
  Cerebral Performance Category (CPC) of 1 to 5. CPC 1: Complete recovery without neurological impairment or conscious with minor impairment. CPC 5: Deceased or brain dead.
Cerebral Performance Category (CPC) after Return of Spontaneous Circulation(ROSC) | Day 90
  Assessment of c-NIRS after Return of Spontaneous Circulation(ROSC) for patients with a good neurological outcome at 90-D. Cerebral Performance Category (CPC) of 1 to 5. CPC 1: Complete recovery without neurological impairment or conscious with minor impairment. CPC 5: Deceased or brain dead
Return of Spontaneous Circulation | 1 hour
  Evaluate the association between the average Cerebral Near infrared spectroscopy (NIRSc) and the occurrence of ROSC (Return of Spontaneous Circulation).
The cumulative dose of adrenaline. | During out-of-hospital cardiopulmonary resuscitation.
  Evaluate the association between the average NIRSc and the cumulative dose of adrenaline (mg/mL)
Resuscitation duration. | During out-of-hospital cardiopulmonary resuscitation.
  Evaluate the association between the average NIRSc and the duration of resuscitation (minutes).
No-flow duration | During out-of-hospital cardiopulmonary resuscitation.
  Evaluate the association between the average NIRSc and the duration of no flow (minutes)
Initial rhythm (Shockable or non-Shockable) | During out-of-hospital cardiopulmonary resuscitation.
  Evaluate the association between the average NIRSc and the inital rhythm (Shockable or non-Shockable)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD-PhD, Study Chair — CHRU de NANCY
Locations (6):
- France (6):
  - CH Colmar- Urgences - SAMU-SMUR, Colmar
  - CHR Metz-Thionville - Mercy hospital -Urgences - SAMU-SMUR, Metz
  - CHRU NANCY - urgences SAMUR SMUR- Central hospital, Nancy
  - CHU Reims - ugences - SAMU-SMUR, Reims
  - Hôpitaux universitaire de Strasbourg - Urgences - SAMU-SMUR, Strasbourg
  - CHR Troyes- Urgences - SAMU-SMUR, Troyes